CLINICAL TRIAL: NCT03332160
Title: A Pilot Study to Evaluate the Feasibility and Potential Effectiveness of the Flexitouch System Head and Neck Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tactile Medical (Industry)
Collaborators: Vanderbilt University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4030
Record Dates: First submitted 2017-10-24; First posted 2017-11-06 (Actual); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Head and Neck Neoplasms; Head and Neck Cancer; Head and Neck Lymphedema
Keywords: Lymphedema; Cancer; Head Cancer; Neck Cancer; Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms; Lymphedema; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of Care (Active Comparator): Standard home lymphedema care
  Interventions: Other: Standard home lymphedema care
- Flexitouch head and neck lymphedema treatment system (Experimental): Daily treatment with Flexitouch® pneumatic compression device for treatment of head and neck lymphedema and standard home lymphedema care
  Interventions: Device: Flexitouch head and neck lymphedema treatment system

INTERVENTIONS:
Device: Flexitouch head and neck lymphedema treatment system — Pneumatic compression device cleared for use by medical professionals and patients who are under medical supervision, for the treatment of many conditions such as: lymphedema; primary lymphedema; post mastectomy edema; edema following trauma and sports injuries; post immobilization edema; venous insufficiency; reducing wound healing time; treatment and assistance in healing stasis dermatitis, venous stasis ulcers, or arterial and diabetic leg ulcers. The Flexitouch system and garments for head and neck are intended for use by medical professionals and patients who are under medical supervision for the treatment of head and neck lymphedema.
  Other Names: Flexitouch System
  Arms: Flexitouch head and neck lymphedema treatment system
Other: Standard home lymphedema care — May include daily self manual lymphatic drainage, exercise, skin care, compression garments (as appropriate).
  Arms: Standard of Care

SUMMARY:
The study will evaluate the feasibility and potential effectiveness of the Flexitouch head and neck treatment plus standard home care compared to standard home care regimen alone.

DETAILED DESCRIPTION:
This study is an open-label, multi-site, stratified randomized, wait list control, pilot study. The study will be conducted at up to 2 sites in the United States and enroll 40 subjects with a diagnosis of head and neck lymphedema following treatment for head and neck cancer. Subjects randomized to receive daily treatment with the Flexitouch pneumatic compression device and home care regimen (SOC) will be seen at baseline and weeks 1, 4, and 8. Subjects randomized to the wait list arm will be seen at baseline and weeks 1, 4, and 8 while receiving SOC treatment. Assessments will include fidelity, satisfaction, symptoms, swelling/inflammation, function, and QOL.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* A previous diagnosis of histologically defined head and neck cancer.
* A diagnosis of head and neck lymphedema.
* Must be able and willing to participate in all aspects of the study and provide informed consent prior to study participation.
* Completed cancer treatment with no evidence of active cancer; all post-surgical swelling must be resolved.
* The head and neck garments must fit appropriately. For patients with a tracheostomy, the fit will be assessed to ensure that the garments do not interfere with their tracheostomy.
* The subject must have experienced at least one of the following:
* Completion of phase 1 lymphedema care in the past 8 weeks;
* The inability to participate/complete phase 1 care due to:
* Lack of available therapist/clinic,
* Lack of insurance coverage or funding to support cost of care.

Exclusion Criteria:

* Uncontrolled hyperthyroidism or parathyroidism (for which endocrinologist recommends against neck compression).
* Carotid sinus hypersensitivity syndrome.
* Symptomatic carotid artery disease, as manifested by a recent transient ischemic attack (within 30 days), ischemic stroke, or amaurosis fugax (monocular visual ischemic symptoms or blindness).
* Symptomatic bradycardia in the absence of a pacemaker.
* Internal jugular venous thrombosis, acute or within 3 months.
* Increased intracranial pressure or other contraindications to internal or external jugular venous compression.
* Acute radiation dermatitis, unhealed surgical scar, unhealed or open wound(s), surgical flap less than 6-8 weeks post-operative.
* Facial or head and neck dermal metastasis.
* Acute facial infection (e.g., facial or parotid gland abscess).
* Any condition in which increased venous and lymphatic return is undesirable.
* History of pulmonary edema or decompensated congestive heart failure with in six (6) week of enrollment.
* Subject is pregnant or trying to become pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-01-02 (Actual); Primary Completion 2019-06-04 (Actual); Study Completion 2019-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Ridner, PhD, RN, Principal Investigator — Vanderbilt University School of Nursing
Locations (2):
- United States (2):
  - SIU School of Medicine, Springfield, Illinois
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Wait-list Control Group: Standard home lymphedema care: May include daily self manual lymphatic drainage (MLD), exercise, skincare, compression garments (as appropriate)
- Interventional Group: Twice daily treatment with Flexitouch® pneumatic compression device and home care regimen, which may include self-MLD exercise, skincare, and wearing an appropriate compression garment, if applicable
Period: Overall Study
Arm/Group | Wait-list Control Group | Interventional Group
Started | 25 | 24
Completed | 24 | 19
Not Completed | 1 | 5
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Developed Exclusion Criteria | 0 | 1
Not completed — Non-adherence to treatment | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Wait-list Control Group: Standard home lymphedema care: May include daily self manual lymphatic drainage, exercise, skincare, compression garments (as appropriate)
- Total: Total of all reporting groups
Arm/Group | Wait-list Control Group | Interventional Group | Total
Number analyzed (Participants) | 24 | 19 | 43
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62.8 [57 to 69] | 61.1 [54 to 68] | 62.2 [56 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 20 | 15 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 24 | 18 | 42
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 24 | 19 | 43
Education [Count of Participants; unit: Participants]
  <=High School | 10 | 6 | 16
  College | 13 | 8 | 21
  Advance Degree | 1 | 5 | 6
Marital Status [Count of Participants; unit: Participants]
  Married/Living with Partner | 20 | 17 | 37
  Other | 4 | 2 | 6
Residence [Count of Participants; unit: Participants]
  City | 8 | 7 | 15
  Country | 12 | 6 | 18
  Suburb | 4 | 6 | 10
Body Mass Index (BMI) at Enrollment [Count of Participants; unit: Participants] — Divided weight (in pounds) by height (in inches) squared and multiplied by 703
  Participants
    Underweight | 1 | 1 | 2
    Normal/Health Weight | 5 | 2 | 7
    Overweight | 10 | 8 | 18
    Obese | 8 | 8 | 16
Smoking history/current [Count of Participants; unit: Participants] | 16 | 12 | 28
Alcohol history/current [Count of Participants; unit: Participants] | 18 | 14 | 32
Tracheotomy at Enrollment [Count of Participants; unit: Participants] | 4 | 2 | 6
Percutaneous Endoscopic Gastrostomy (PEG) at Enrollment [Count of Participants; unit: Participants] | 6 | 6 | 12
Months since Lymphedema Diagnosis [Median (Inter-Quartile Range); unit: months] | 5.3 [1 to 10] | 5.2 [1 to 18] | 5.2 [1 to 14]
Months since Initial Lymphedema Treatment [Median (Inter-Quartile Range); unit: months] | 4.6 [2 to 9] | 4.5 [2 to 22] | 4.6 [2 to 12]

OUTCOME MEASURES:

1. Primary Outcome: Fidelity/Adherence Via Subject Diary
Description: Evaluate the feasibility and potential effectiveness of the Flexitouch head and neck garments by monitoring fidelity/adherence using a subject diary. Values represent a count of participants who met the prescribed use criteria by week. The prescribed use was defined as two 30 minute sessions in a day.
Time Frame: From baseline to end of treatment at 8 weeks
Population: This analysis only applies to the Interventional Group.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Group
Number analyzed (Participants) | 19
Participants
  Week 1: 0 days | 5
  Week 1: 1 day | 1
  Week 1: 2 days | 1
  Week 1: 3 days | 2
  Week 1: 4 days | 1
  Week 1: 5 days | 3
  Week 1: 6 days | 1
  Week 1: 7 days | 5
  Week 2: 0 days | 4
  Week 2: 1 day | 1
  Week 2: 2 days | 0
  Week 2: 3 days | 1
  Week 2: 4 days | 4
  Week 2: 5 days | 3
  Week 2: 6 days | 1
  Week 2: 7 days | 5
  Week 3: 0 days | 4
  Week 3: 1 day | 0
  Week 3: 2 days | 1
  Week 3: 3 days | 2
  Week 3: 4 days | 2
  Week 3: 5 days | 4
  Week 3: 6 days | 2
  Week 3: 7 days | 4
  Week 4: 0 days | 3
  Week 4: 1 day | 1
  Week 4: 2 days | 3
  Week 4: 3 days | 2
  Week 4: 4 days | 2
  Week 4: 5 days | 2
  Week 4: 6 days | 3
  Week 4: 7 days | 3
  Week 5: 0 days | 4
  Week 5: 1 day | 2
  Week 5: 2 days | 2
  Week 5: 3 days | 0
  Week 5: 4 days | 2
  Week 5: 5 days | 5
  Week 5: 6 days | 1
  Week 5: 7 days | 3
  Week 6: 0 days | 2
  Week 6: 1 day | 2
  Week 6: 2 days | 0
  Week 6: 3 days | 2
  Week 6: 4 days | 4
  Week 6: 5 days | 3
  Week 6: 6 days | 2
  Week 6: 7 days | 4
  Week 7: 0 days | 3
  Week 7: 1 day | 1
  Week 7: 2 days | 2
  Week 7: 3 days | 3
  Week 7: 4 days | 1
  Week 7: 5 days | 2
  Week 7: 6 days | 2
  Week 7: 7 days | 5
  Week 8: 0 days | 4
  Week 8: 1 day | 2
  Week 8: 2 days | 3
  Week 8: 3 days | 2
  Week 8: 4 days | 4
  Week 8: 5 days | 1
  Week 8: 6 days | 2
  Week 8: 7 days | 1

2. Primary Outcome: Adverse Events
Description: Evaluate the feasibility and potential effectiveness of the Flexitouch head and neck garments by monitoring adverse events using the CTCAE (v4.0). Values represent the count of events per adverse events category.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Number; unit: Events
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
Events
  Cardiac disorders | 3 | 0
  Ear and labyrinth disorders | 1 | 1
  Endocrine disorders | 2 | 2
  Eye disorders | 1 | 0
  Gastrointestinal disorders | 3 | 3
  General disorders | 7 | 2
  Immune system disorders | 1 | 0
  Infections and infestations | 7 | 1
  Musculoskeletal and connective tissue disorders | 0 | 2
  Neoplasms benign, malignant and unspecified | 1 | 0
  Nervous system disorders | 6 | 7
  Psychiatric disorders | 2 | 0
  Skin and subcutaneous tissue disorders | 5 | 1
  Surgical and medical procedures | 1 | 3
  Respiratory, thoracic and mediastinal disorders | 10 | 5
  Vascular disorders | 3 | 1

3. Primary Outcome: Treatment Satisfaction
Description: Evaluate the feasibility and potential effectiveness of the Flexitouch head and neck garments by monitoring treatment satisfaction using a satisfaction survey. A survey assessed participants' perceived ability to control their head and neck lymphedema before (at baseline) and after the usage of the Flexitouch at 8 weeks. Values represent a count of participants who indicated good, very good, or excellent.
Time Frame: From baseline to the end of treatment at 8 weeks
Population: This only applied to participants in the interventional group who had indicated good, very good, or excellent in regards to their perceived ability to control their head and neck lymphedema.
Measure: Count of Participants; unit: Participants
Arm/Group | Interventional Group
Number analyzed (Participants) | 19
Participants
  Baseline (Good, Very Good, or Excellent) | 5
  8 Weeks (Good, Very Good, or Excellent) | 16

4. Secondary Outcome: Reduction in Swelling/Inflammation - Endoscopy
Description: The change in percent of sites with visible swelling and inflammation as assessed via endoscopy (using Modified Patterson Scale) from baseline to week 8. The range for each anatomical structure includes 1-4: Normal, Mild, Moderate, and Severe. A lower score means a better outcome. A greater negative value indicates a greater reduction in swelling. Total score range: 0-100%.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Median (Inter-Quartile Range); unit: Change in score
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
Change in score | -2.7778 [-16.6667 to 5.5556] | -11.1111 [-31.3725 to 8.0882]

5. Secondary Outcome: Reduction in Swelling/Inflammation - Cytokine Levels
Description: The presence of swelling and inflammation was assessed in all participants via the change in cytokine levels of Interleukin 6 (IL-6) at baseline to week 8. A lower score means a better outcome. A greater negative value indicates a greater reduction in cytokine levels.
Time Frame: From baseline to the end of treatment at 8 weeks
Population: Not all participants' blood samples were analyzable.
Measure: Median (Inter-Quartile Range); unit: fg/ml
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 20 | 18
fg/ml | -836.47 [-8411.52 to 1142.85] | -275.68 [-3772.13 to 4367.30]

6. Secondary Outcome: Reduction in Swelling/Inflammation - Digital Photography
Description: The presence of swelling and inflammation was assessed in all participants by digital photography at baseline and 8 weeks. A lower value means a better outcome. A greater negative value indicates a greater reduction in swelling. Three views were scored each with 30 grids. The percentage of views with visible swelling was determined. The score ranged from 0-100%.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
score on a scale
  Front View Change | 4.924 [-11.601 to 12.064] | -24.308 [-29.167 to -7.143]
  Right View Change | -7.279 [-13.991 to 2.143] | -22.368 [-27.273 to -14.286]
  Left View Change | -4.4466 [-17.2348 to 6.8062] | -16.5217 [-21.7391 to -2.3810]

7. Secondary Outcome: Reduction in Swelling/Inflammation - Grading of External Lymphedema
Description: The presence of swelling and inflammation was assessed in all participants through grading of external lymphedema via the Head and Neck Lymphedema and Fibrosis Assessment criteria (HNLEF) during a physical examination at baseline and 8 weeks. A total of 9 sites were evaluated for the presence of lymphedema and graded from 1 (mild) to 3 (severe) at each site. The number of sites ranged from 0-9 with a total severity score ranging from 0-27. Results are the change in a total score between baseline and 8 weeks. A lower score indicates a better outcome. A greater negative value indicates a greater reduction in swelling.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
score on a scale | -0.5000 [-1.0000 to 2.0000] | 0.0000 [-6.0000 to 2.0000]

8. Secondary Outcome: Function - Jaw Range of Motion
Description: The function was assessed in all participants at baseline and week 8 through the jaw range of motion measurements using the Therabite Jaw ROM Scale. The TheraBite Jaw ROM Scale was used to measure in millimeters the jaw opening of the maximum inter-incisal distance (upper right central to lower right central incisor). The values were categorized by grade change. The change of -1 indicates the severity improved by one grade. A value of zero indicates a participant remained stable. A value of 1 indicates a patient worsened by one grade.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
Participants
  -1 | 4 | 1
  0 | 18 | 17
  1 | 2 | 1

9. Secondary Outcome: Function - Neck Disability Index
Description: The function was assessed in all participants at baseline and week 8 by the Neck Disability Index (NDI). Values represent a change from baseline. Minimum score: 0 with a minimum disability of 0%. Maximum score: 50 with a maximal disability of 100%.
  0 - 20% (minimal) - The patient can cope with most living activities. Usually, no treatment is indicated apart from advice on lifting sitting and exercise.
  21 - 40% (moderate) - The patient experiences more pain and difficulty with sitting lifting and standing. Travel and social life are more difficult and they may be disabled from work. The patient can usually be managed by conservative means.
  41 - 60% (severe) -Pain remains the main problem in this group but activities of daily living are affected. These patients require a detailed investigation.
  61 - 80% (crippled) - Pain impinges on all aspects of the patient's life. Positive intervention is required.
  81 - 100% (bed bound) - Need to exclude exaggeration or malingering.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
score on a scale | 1.00 [-4.00 to 9.50] | 0.00 [-4.00 to 0.00]

10. Secondary Outcome: Function - Voice Handicap Index
Description: The function was assessed in all participants at baseline and week 8 by the Voice Handicap Index (VHI). Values represent a change from baseline. Max / Min Total Score: 0-120. A lower score indicates a better outcome.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
score on a scale | 0.50 [-1.94 to 2.75] | 0.00 [-3.00 to 3.00]

11. Secondary Outcome: Function - Cervical and Shoulder Range of Motion
Description: The function was assessed in all participants at baseline and week 8 through the cervical range of motion (CROM) and shoulder range of motion (SROM) measurements. A positive value indicates a better outcome. The greater the value, the greater the change from baseline.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Median (Inter-Quartile Range); unit: Degrees
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
Degrees
  CROM Forward Flexion | -1.00 [-8.75 to 8.50] | -2.00 [-5.00 to 2.00]
  CROM Extension | 4.00 [-5.75 to 12.75] | 1.00 [-6.00 to 6.00]
  CROM Left Lateral Rotation | -1.00 [-6.50 to 3.00] | -1.00 [-6.00 to 6.00]
  CROM Right Lateral Rotation | -0.50 [-7.00 to 3.50] | 1.00 [-8.00 to 5.00]
  SROM Forward Flexion (Right Active) | 0.00 [-3.50 to 6.75] | 1.50 [-1.00 to 11.00]
  SROM Forward Flexion (Left Active) | -0.75 [-6.37 to 9.13] | 7.50 [-1.50 to 9.50]
  SROM Abduction (Right Active) | 7.00 [-9.00 to 17.00] | 3.00 [0.00 to 13.00]
  SROM Abduction (Left Active) | 5.50 [-13.12 to 12.88] | 5.00 [-5.50 to 15.00]
  SROM External Rotation (Right Active) | -1.25 [-8.87 to 5.00] | 0.00 [-8.00 to 4.00]
  SROM External Rotation (Left Active) | -2.25 [-6.50 to 1.88] | 2.50 [-1.00 to 6.50]

12. Secondary Outcome: Symptoms - Vanderbilt Head and Neck Symptom Survey
Description: Symptoms were assessed in all participants at baseline and week 8 via the Vanderbilt Head and Neck Symptom Survey plus General Symptom Survey (VHNSS v2.0 plus GSS). Values represent a median score change from baseline. Score range: 0-10. A lower score indicates a better outcome. A more negative value indicates a greater change from baseline. Given this was a self-reported survey, responses were not mandatory and thus missing for some subjects.
Time Frame: From baseline to the end of treatment at 8 weeks
Population: Data was not available and/or applicable to all participants in certain categories.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
score on a scale
  Mouth Pain | 0.00 [-1.29 to 0.50] | 0.00 [-1.50 to 0.00]
  General Pain | 0.67 [-0.25 to 2.08] | 0.00 [-1.33 to 0.00]
  Swallowing Solids: number analyzed (Participants) | 22 | 16
  Swallowing Solids | -0.06 [-1.12 to 0.73] | -0.25 [-2.25 to 0.00]
  Swallowing Liquids: number analyzed (Participants) | 23 | 18
  Swallowing Liquids | 0.00 [-1.00 to 1.00] | 0.00 [-.12 to 0.00]
  Nutrition | 0.00 [-0.94 to 1.13] | 0.00 [-1.00 to 0.25]
  Mucous | -0.12 [-0.75 to 0.69] | -0.50 [-1.75 to 0.00]
  Dry Mouth | 0.20 [-0.55 to 0.90] | 0.00 [-0.20 to 0.40]
  Taste/Smell: number analyzed (Participants) | 22 | 17
  Taste/Smell | -0.25 [-1.83 to 0.71] | -0.17 [-1.42 to 0.45]
  Voice | -0.67 [-1.33 to 0.25] | -.033 [-0.67 to 1.00]
  Teeth: number analyzed (Participants) | 17 | 18
  Teeth | 0.25 [0.00 to 1.13] | 0.00 [0.00 to 0.54]

13. Secondary Outcome: Quality of Life - Linear Analog Self-Assessment
Description: Quality of life was assessed in all participants at baseline and week 8 using the Linear Analog Self-Assessment. The total score for the assessment ranged from 0-50. Each category represents a change in score from the baseline visit which ranged from positive 4 to negative 4. A positive change indicates an improvement. Values represent the count of participants in each category.
Time Frame: From baseline to the end of treatment at 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
Participants
  -4 | 1 | 0
  -2 | 1 | 0
  -1 | 5 | 3
  0 | 10 | 13
  1 | 4 | 2
  2 | 2 | 1
  4 | 1 | 0

14. Secondary Outcome: Symptoms - Lymphedema Symptom Intensity and Distress Survey
Description: Lymphedema Symptom Intensity and Distress Survey-Head and Neck (LSIDS-HN) assessed the measurement characteristics of a symptom burden for participants with head and neck lymphedema at baseline and week 8. Each symptom was rated on intensity and distress using a 5-point scale. A maximum response for any symptom within a given cluster was used for the analysis. The total score ranged from 0-10. The values represent a change from baseline. A lower score means a better outcome.
Time Frame: From baseline to the end of treatment at 8 weeks
Population: Data may be missing or left blank by participant.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Wait-list Control Group | Interventional Group
Number analyzed (Participants) | 24 | 19
score on a scale
  Soft Tissue | 0.00 [0.00 to 2.00] | -2.00 [-2.00 to 0.00]
  Neurological | 0.00 [0.00 to 2.00] | 0.00 [-2.00 to 0.00]
  Oral | 0.00 [-1.00 to 2.00] | 0.00 [-2.00 to 0.00]
  BioBehavioral | 0.00 [-1.75 to 0.75] | 0.00 [-2.00 to 1.00]
  Resources | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  Sexuality: number analyzed (Participants) | 23 | 19
  Sexuality | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.00]
  Activity | 0.00 [-2.75 to 1.00] | 0.0 [-3.00 to 0.00]
  Function | 0.00 [-0.75 to 2.00] | 0.00 [-1.00 to 1.00]

ADVERSE EVENTS:
Time Frame: 8 weeks; and an additional 8 weeks for the Wait-List Control participants who participated in the optional follow-up period.
Arm/Group | Wait-list Control Group | Interventional Group
All-Cause Mortality (participants affected / at risk) | 1/24 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/24 | 2/19
Other Adverse Events (participants affected / at risk) | 20/24 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wait-list Control Group (N=24) | Interventional Group (N=19)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Sudden death NOS (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Wait-list Control Group (N=24) | Interventional Group (N=19)
Chest Pain - Cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Hypertension (Cardiac disorders) | 1 (2) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Corneal ulcer (Eye disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Aphonia (General disorders) | 1 (1) | 0 (0)
General disorders and administration site conditions - other specify (General disorders) | 1 (1) | 0 (0)
Neck pain (General disorders) | 1 (1) | 1 (1)
Oral pain (General disorders) | 1 (1) | 1 (1)
Pain (General disorders) | 3 (3) | 1 (1)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Middle ear inflammation (Infections and infestations) | 1 (1) | 1 (1)
Pneumonitis (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 2 (3) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 2 (4)
Myelitis (Nervous system disorders) | 1 (1) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2) | 0 (0)
Spasiticity (Nervous system disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin infection (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 (1) | 3 (3)
Infection and infestation - Other, specify (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This trial was designed as a pilot study and thus the sample size is small.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Informed Consent Form (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/60/NCT03332160/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-09-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03332160/Prot_SAP_001.pdf